CLINICAL TRIAL: NCT00252850
Title: A Phase I, Open-Label Study of CERE-120 (Adeno-Associated Virus Serotype 2 [AAV2]-Neurturin[NTN] to Assess the Safety and Tolerability of Intrastriatal Delivery to Subjects With Idiopathic Parkinson's Disease
Brief Title: Safety of CERE-120 (AAV2-NTN) in Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Ceregene (Industry)
Responsible Party: Joao Siffert, Chief Medical Officer, Ceregene
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERE-120-01
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2016-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Gene Transfer
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: CERE-120: AAV2-NTN

SUMMARY:
This is a Phase I dose escalating open-label study designed to assess the safety, tolerability and biologic activity of an in vivo AAV2 mediated delivery of the gene encoding NTN (CERE-120).

Twelve (up to 18) subjects will receive one of two open-label doses of CERE-120 via bilateral stereotactic injections targeting the putaminal region of the brain. Subjects will be enrolled in one of two cohorts, a low-dose cohort of six subjects followed by a high dose cohort of six subjects.

The design of this study is such that the primary objective, the evaluation of safety and tolerability, will be assessed by frequent observations for adverse events, clinical laboratory test results, imaging (MRI), neuropsychometric testing, and evaluations of disease status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral idiopathic Parkinson's Disease of at least 5 years duration since diagnosis with motor fluctuations, despite adequate oral antiparkinsonian therapy.
* Diagnosis of moderate to severe Parkinson's Disease based on clinical rating scales.
* Males or nonpregnant females 35-75 years of age, inclusive.
* Stable medication requirements, and clear response to antiparkinsonian medications during the 60-day eligibility evaluation period.
* No conditions that would render the subject unsuitable for surgery, or that would interfere with any of the assessments of safety or efficacy in this trial.
* Subject's informed consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* A history of any clinically significant medical, psychiatric, or laboratory abnormality for which participation in the study would pose a safety risk to the subject.
* History of treatment of Parkinson's disease by any procedure involving intracranial surgery or implantation of a device.
* MRI of the brain within 12 months before the anticipated dosing procedure that indicates the presence of an abnormality that may interfere with the assessments of safety or efficacy or would, in the judgment of the investigator, present a surgical risk to the subject.
* Any disorder that precludes a surgical procedure or alters wound healing.
* A score of less than or equal to 25 on the Folstein Mini-Mental examination performed during the eligibility evaluation period.
* Chemotherapy, cytotoxic therapy, or immunotherapy within 6 weeks prior to CERE-120 administration.
* Vaccinations within 30 days prior to CERE-120 administration.
* History, within two years before the anticipated dosing procedure, of drug or alcohol abuse.
* Treatment with nonantiparkinsonian agents that may affect symptoms of Parkinson's disease within 60 days before the anticipated dosing procedure.
* Any medical disability that would interfere with the assessment of safety and efficacy in this trial or would compromise the ability of the subject to undergo study procedures (e.g. MRI, PET) or to give informed consent.
* History of prior gene transfer therapy.
* Treatment with an investigational agent within 60 days before the anticipated dosing procedure.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Marks, Jr., M.D., Principal Investigator — University of California, San Francisco; Leo Verhagen Metman, M.D., Ph.D., Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois

REFERENCES:
- [Result] Marks WJ Jr, Ostrem JL, Verhagen L, Starr PA, Larson PS, Bakay RA, Taylor R, Cahn-Weiner DA, Stoessl AJ, Olanow CW, Bartus RT. Safety and tolerability of intraputaminal delivery of CERE-120 (adeno-associated virus serotype 2-neurturin) to patients with idiopathic Parkinson's disease: an open-label, phase I trial. Lancet Neurol. 2008 May;7(5):400-8. doi: 10.1016/S1474-4422(08)70065-6. Epub 2008 Apr 2. PMID 18387850